CLINICAL TRIAL: NCT05933460
Title: Investigation of the Impact of the Administration of Crocus Sativus L Extract on the Metabolic Control of Patients With Type 1 Diabetes Mellitus
Brief Title: Crocus Sativus Extract Impact in Metabolic Control of Patients With Diabetes Mellitus Type 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Prof. Triantafyllos Didangelos, Professor of Internal Medicine- Diabetology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Diabetes1Crocus; 1.46-21/11/2018 (Other: Aristotle University of Thessaloniki)
Record Dates: First submitted 2023-05-14; First posted 2023-07-06 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes type1
Keywords: diabetes mellitus type 1; diabetes type 1; saffron; saffron extract; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Dietary Supplements; Probiotics; Prebiotics; Magnesium

STUDY DESIGN:
Intervention Model Description: Double blind placebo controlled randomized trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: No participant or personnel knew the randomization process and the only knew did not had to do with participants or administration of supplement or collecting data. The company providing the supplement did not know either.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Group (Experimental): A sachet of a combination of 4 strains of probiotics (1billion CFU) (Lactobacillus rhamnosus, Bifidobacterium animalis lactis, Bifidobacterium breve, Bifidobacterium longum), Fructooligosaccharides 100mg, Magnesium 75mg and Crocus sativus (Saffron extract 28mg) was administered 3 times per day in people with diabetes type 1 for 6 months on continuous glucose monitoring systems.
  Interventions: Dietary Supplement: dietary supplement with probiotics, prebiotics, magnesium and saffron extract
- Placebo group (Placebo Comparator): A sachet of a combination of 4 strains of probiotics (1billion CFU(Lactobacillus rhamnosus, Bifidobacterium animalis lactis, Bifidobacterium breve, Bifidobacterium longum), Fructooligosaccharides 100mg, Magnesium 75mg without crocus sativus was administered 3 times per day in people with diabetes type 1 for 6 months on continuous glucose monitoring systems.
  Interventions: Dietary Supplement: dietary supplement with probiotics, prebiotics, magnesium

INTERVENTIONS:
Dietary Supplement: dietary supplement with probiotics, prebiotics, magnesium and saffron extract — A sachet of a combination of 4 strains of probiotics (1billion CFU) (Lactobacillus rhamnosus, Bifidobacterium animalis subscp. lactis, Bifidobacterium breve, Bifidobacterium longum), Fructooligosaccharides 100mg, Magnesium 75mg and Saffron extract 28mg was administered 3 times per day
  Other Names: Probiotics and saffron extract
  Arms: Active Group
Dietary Supplement: dietary supplement with probiotics, prebiotics, magnesium — A sachet of a combination of 4 strains of probiotics (1billion CFU) (Lactobacillus rhamnosus, Bifidobacterium animalis subscp. lactis, Bifidobacterium breve, Bifidobacterium longum), Fructooligosaccharides 100mg, Magnesium 75mg was administered 3 times per day
  Other Names: Probiotics
  Arms: Placebo group

SUMMARY:
Administration of 4 strain of probiotics, prebiotic, magnesium and crocus sativus extract in a sachet to people with diabetes mellitus type 1 for 6 months

DETAILED DESCRIPTION:
Double blind placebo controlled randomized trial: A sachet of a combination of 4 strains of probiotics (Lactobacillus rhamnosus, Bifidobacterium animalis lactis, Bifidobacterium breve, Bifidobacterium longum), Fructooligosaccharides, Magnesium and Saffron extract was administered 3 times per day in people with diabetes type 1 for 6 months on continuous glucose monitoring systems.

ELIGIBILITY:
Inclusion Criteria:

* People with diabetes mellitus type 1 (with diabetes duration over 1 year) (adults <18 years old) wearing a continuous glucose monitoring system with or without an insulin pump

Exclusion Criteria:

* Pregnant
* People with diabetes mellitus type 2
* Breastfeeding women
* People with liver disease
* People with chronic kidney disease (over stage 3)
* People with allergy in crocus sativus
* People that consume everyday herbs or supplements
* People on anti platelet treatment not for prevention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
glycated hemoglobin | 6 months
  glycated hemoglobin %
blood glucose | 6 months
  Fasting blood glucose (mg/dl)
serum cholesterol | 6 months
  Total Cholesterol mg/dl
serum High density lipoprotein cholesterol | 6 months
  High density lipoprotein Cholesterol mg/dl
serum low density lipoprotein cholesterol | 6 months
  Low density lipoprotein cholesterol mg/dl
triglycerides | 6 months
  serum Triglycerides mg/dl
Systolic Blood pressure | 6 months
  Systolic blood pressure mmHg
Diastolic Blood pressure | 6 months
  Diastolic blood pressure mmHg

SECONDARY OUTCOMES:
Continuous glucose monitoring data | 6 months
  Time in range %
Continuous glucose monitoring time | 6 months
  Time below range %
Continuous glucose monitoring time data | 6 months
  Time above range %
Continuous glucose monitoring glycemic data | 6 months
  Glucose Management Indicator %
Continuous glucose monitoring statistic data | 6 months
  Coefficient of variance
Sural nerve conduction velocity | 6 months
  Nerve conduction velocity is measured in the sural sensory nerve of both feet with Neurometrix DPNCheck
Electrochemical skin conductance | 6 months
  Sudomotor function was assessed with SUDOSCAN, which measures electrochemical skin conductance in the feet (ESCF) and hands (ESCH)
Cardiovascular Autonomic Reflex tests | 6 months
  Autonomic neuropathy testing included cardiovascular autonomic reflex tests (CARTs) such as heart rate variability to obtain mean circular resultant (MCR), and the 30:15 stand up test to obtain postural index and blood pressure measurement to test for orthostatic hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Triantafyllos Didangelos, Professor, Study Director — Aristotle University Of Thessaloniki
Locations (1):
- University General Hospital of Thessaloniki AHEPA, Thessaloniki, Central Macedonia, Greece

IPD SHARING:
Plan to Share IPD: No
There is no plan for sharing individual participant data due to bioethics committee restrictions on personal data privacy

REFERENCES:
- [Background] Giannoulaki P, Kotzakioulafi E, Chourdakis M, Hatzitolios A, Didangelos T. Impact of Crocus Sativus L. on Metabolic Profile in Patients with Diabetes Mellitus or Metabolic Syndrome: A Systematic Review. Nutrients. 2020 May 14;12(5):1424. doi: 10.3390/nu12051424. PMID 32423173